CLINICAL TRIAL: NCT05311839
Title: Combined Effect of Graded Thera Band and Scapular Stabilization Exercises on Shoulder Adhesive Capsulitis Post Mastectomy
Brief Title: Effect of Thera Band Exercises on Adhesive Capsulitis Post Mastectomy
Acronym: Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maged Basha (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah. Consultant Physical Therapist, El-Sahel Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Cairo, Egypt., Qassim University
Organization: Qassim University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT3465
Record Dates: First submitted 2022-03-26; First posted 2022-04-05 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thera band exercises group (Experimental): received graded Thera band exercises for 5 days per week for eight weeks in addition to the conventional physical therapy program.
  Interventions: Other: Exercise; Other: Thera band
- conventional physiotherapy program group (Experimental): received a conventional physical therapy program.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Hot packs, active range of motion exercises, pendular exercises, wall climb exercises, mobilization exercises, and shoulder capsular stretching
  Other Names: conventional physical therapy program
Other: Thera band — graded Thera band exercises for shoulder flexion, abduction, internal, and external rotation
  Other Names: graded Thera band exercises and scapular stabilization exercises
  Arms: Thera band exercises group

SUMMARY:
Breast cancer surgeries particularly mastectomy results in limited shoulder movement which can lead to arm, shoulder pain and stiffness. Females who underwent mastectomy have reported a significantly higher incidence of shoulder morbidity

DETAILED DESCRIPTION:
Exercise therapy might help in reduction of pain and restoration of the range, coordination and control of movement in patients with adhesive capsulitis. Graded resistance exercises are effective in decreasing fatigue levels, enhancing functional capacity and muscle strength. Rehabilitation exercises which strengthen the scapular stability can be extremely beneficial in rehabilitation treatment of patients with shoulder pain and problems

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 40-60 years.
* 2nd stage of adhesive capsulitis,
* Shoulder pain and stiffness for at least 3 months.
* Restriction in shoulder flexion, abduction, internal and external rotation ROM less than 50% when compared to the other shoulder.

Exclusion Criteria:

* Shoulder or acromioclavicular joint osteoarthritis.
* Bone diseases.
* Infection.
* Severe osteoporosis.
* Tumors or metastasis.
* History of previous shoulder trauma or accidental injuries.
* Previous history of dislocation.
* Previous history of surgery on the specific shoulder.
* Any other shoulder problems.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breast Cancer, post-mastectomy
Enrollment: 70 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Shoulder range of motion | at baseline
  A digital goniometer flexion and abduction, internal and external rotation range of motion
Shoulder range of motion | after 8 weeks
  A digital goniometer flexion and abduction, internal and external rotation range of motion
physical function | at baseline
  the Disability of the Arm, Shoulder, and Hand questionnaire [DASH] is used to measure physical function
physical function | after 8weeks
  the Disability of the Arm, Shoulder, and Hand questionnaire [DASH] is used to measure physical function
Health-related quality of life | at baseline
  assessed using the Medical Outcomes Study short-form (SF-36).
Health-related quality of life | after 8 weeks
  assessed using the Medical Outcomes Study short-form (SF-36).

SECONDARY OUTCOMES:
Muscle strength | at baseline
  A handheld dynamometer (J Tech Commender Muscle Tester, Salt Lake City, Utah, USA)
Muscle strength | after 8 weeks
  A handheld dynamometer (J Tech Commender Muscle Tester, Salt Lake City, Utah, USA)
Visual analogue scale | at baseline
  used to assess the intensity of shoulder pain. consists of 10-cm line, and was utilized to quantify the pain severity within shoulder, where the score of zero means no pain, while a score of ten means significant pain
Visual analogue scale | after 8 weeks
  used to assess the intensity of shoulder pain.consists of 10-cm line, and was utilized to quantify the pain severity within shoulder, where the score of zero means no pain, while a score of ten means significant pain

CONTACTS AND LOCATIONS:
Overall Officials: Noha Kamel, PhD, Principal Investigator — Cairo University; Nancy Aboelnour, PhD, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Cheing GL, So EM, Chao CY. Effectiveness of electroacupuncture and interferential eloctrotherapy in the management of frozen shoulder. J Rehabil Med. 2008 Mar;40(3):166-70. doi: 10.2340/16501977-0142. PMID 18292916
- [Result] Dilaveri CA, Sandhu NP, Neal L, Neben-Wittich MA, Hieken TJ, Mac Bride MB, Wahner-Roedler DL, Ghosh K. Medical factors influencing decision making regarding radiation therapy for breast cancer. Int J Womens Health. 2014 Nov 19;6:945-54. doi: 10.2147/IJWH.S71591. eCollection 2014. PMID 25429241
- [Result] Sabari JS, Maltzev I, Lubarsky D, Liszkay E, Homel P. Goniometric assessment of shoulder range of motion: comparison of testing in supine and sitting positions. Arch Phys Med Rehabil. 1998 Jun;79(6):647-51. doi: 10.1016/s0003-9993(98)90038-7. PMID 9630143
- [Derived] Aboelnour NH, Kamel FH, Basha MA, Azab AR, Hewidy IM, Ezzat M, Kamel NM. Combined effect of graded Thera-Band and scapular stabilization exercises on shoulder adhesive capsulitis post-mastectomy. Support Care Cancer. 2023 Mar 16;31(4):215. doi: 10.1007/s00520-023-07641-6. PMID 36922413